CLINICAL TRIAL: NCT04850560
Title: Sequential Low-dose Decitabine Therapy With Novel CAR-T Carrying PD-1/CD28 Chimeric Switch Receptor in Relapsed or Refractory B-cell Lymphoma
Brief Title: Sequential Low-dose Decitabine With PD-1/CD28 CD19 CAR-T in Relapsed or Refractory B-cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR2021001123
Record Dates: First submitted 2021-04-18; First posted 2021-04-20 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-04

CONDITIONS: Objective Response Rate
MeSH Terms: interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19 PD-1/CD28 CAR-T Plus Low Dose Decitabine (Experimental)
  Interventions: Biological: CD19 PD-1/CD28 CAR-T Plus Low Dose Decitabine

INTERVENTIONS:
Biological: CD19 PD-1/CD28 CAR-T Plus Low Dose Decitabine — CD19 PD-1/CD28 CAR-T Plus Low Dose Decitabine

SUMMARY:
To evaluate the efficacy and safety of CD19 PD-1/CD28-CAR-T sequential low-dose decitabine in the treatment of relapse or refractory B cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥ 18, upper limit 75, unlimited for men and women;

  (2) ECOG score 0-3;

  (3) Histologically confirmed diffuse large B-cell lymphoma (DLBCL) [according to who 2008];

  (4) CD19 was positive (immunohistochemistry or flow cytometry).

  (5) The definition of refractory or relapse of DLBCL is: no complete remission after 2-line treatment; disease progression in any treatment process, or disease stabilization time equal to or less than 6 months; or disease progression or relapse within 12 months after hematopoietic stem cell transplantation;

  (6) The previous treatment of diffuse large B cell lymphoma must include rituximab (CD20 mAb) and anthracycline;

  (7) There should be at least one measurable focus. It is required that any length of lymph node focus should be greater than 1.5cm or any length of extranodal focus should be greater than 1.0cm. PET-CT scan focuses should have uptake (SUV is greater than liver blood pool);

  (8) The absolute value of neutrophils in peripheral blood ≥ 1000 / μ L, platelet ≥ 45000 / μ L;

  (9) Heart, liver and kidney function: creatinine < 1.5mg/dl; ALT (alanine aminotransferase) / AST (aspartate aminotransferase) 2.5 times lower than the normal upper limit; total bilirubin < 1.5mg/dl; heart ejection fraction (EF) ≥ 50%;

  (10) Sufficient understanding ability and voluntary signing of informed consent;

  (11) Those with fertility must be willing to use contraceptive methods;

  (12) According to the judgment of the researchers, the expected survival time is more than 4 months;

  (13) Willing to follow visit schedule, administration plan, laboratory inspection and other test steps.

Exclusion Criteria:

* (1) History of other tumors;

  (2) Hematopoietic stem cell transplantation was performed within 6 weeks;

  (3) Any target car-t treatment was performed within 3 months before the car-t treatment;

  (4) Previous use of any commercially available PD-1 mAb;

  (5) Cytotoxic drugs, glucocorticoids and other targeted drugs were received within 2 weeks before cell collection;

  (6) Active autoimmune diseases;

  (7) Uncontrollable infection of active bacteria and fungi;

  (8) HIV infection, syphilis infection; active hepatitis B or C: hepatitis B: HBV-DNA ≥ 1000IU / ml; hepatitis C: HCV RNA positive and liver function abnormal.

  (9) Known central nervous system lymphoma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 3 months
  Objective response rate of the combination

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No